CLINICAL TRIAL: NCT00613288
Title: Testosterone and Lipolysis, Insulin Sensitivity and Protein Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: MD, PhD, DMSc Claus H. Gravholt, Medical Departmnt M, Endocrinology and Diabetes, Aarus University Hospital, NBG
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: M-20070046
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Hypogonadism
Keywords: acute; testosterone; experimental; hypogonadism; lipolysis; insulin sensitivity; protein; metabolism; Experimental hypogonadism; Testosterone substitution
MeSH Terms: conditions — Hypogonadism; Insulin Resistance | interventions — Testosterone; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Testosterone (Testogel), GnRH analog (Leuprorelide) and Placebo

INTERVENTIONS:
Drug: Testosterone (Testogel), GnRH analog (Leuprorelide) and Placebo — The trial is a double blinded, randomised cross-over study of 4 x 2 days with an interval of 1 month in between. 12 healthy young male participants will receive the GnRH-agonist leuprorelide 7,5 mg s.c. 3 weeks before examination on 3 occasions, and a fourth day without intervention.
  The four days will include treatment on the examination day, Day 1 with:
  1. Placebo (hypogonadism after leuprorelide injection)
  2. Testosterone gel 50 mg applicated in the morning at 06.00 am (physiologic substitution - after leuprorelide injection).
  3. Testosterone gel 150 mg applicated in the morning at 06.00 am (supra-physiologic substitution - after leuprorelide injection).
  4. No treatment.

SUMMARY:
Testosterone(T) has known effects on many organ systems, although many of its metabolic actions are unrevealed. T is an anabolic hormone stimulating protein synthesis but this effect has barely been investigated in controlled studies. It also has lipolytic actions influencing body composition, but little is known of its regional impact on fat tissue. T affects insulin sensitivity. There is an increased incidence of hypogonadism in type 2 diabetes, and among patients with hypogonadism there is an increased incidence of type 2 diabetes. The actions of testosterone on glucose metabolism are unknown.

The purpose of this study is therefore to:

Investigate the lipolytic effect of testosterone on muscle and fat tissue. To gain insight in the intracellular mechanisms of testosterone on lipolysis and investigate possible regional differences in lipolysis and changes in body composition.

Finally to investigate the effect of short term experimental hypogonadism and acute testosterone substitution on cytokines, insulin sensitivity and protein metabolism.

The trial is a randomised double blinded cross-over study of 4 x 2 days with an interval of 1 month in between. 12 healthy young men will receive GnRH treatment over a 3 month period and examined on 4 occasions with various degrees of T substitution and placebo . The examinations take place at the Research Lab within the Medical Department M.

The investigations are deemed relevant to the understanding of the interrelationship between male hypogonadism and type 2 diabetes. The hypothesis is that T has beneficial effects on carbohydrate, fat and protein metabolism. The generated knowledge would therefore hopefully improve prophylaxis, screening and early treatment of both group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 20-35
* Normal biochemical screen and ECG

Exclusion Criteria:

* Heart disease
* BMI>25
* Diabetes
* Antecedent or present cancer
* Vascular disease
* Antecedent or present hormone treatment
* Medical treatment with known effects on fat metabolism
* Big X-ray examinations equivalent to, or more than a chest x-ray and all kinds of CT scans until 6 month before the start of the study and during the study.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Testosterone influence on Insulin Sensitivity, Lipolysis and protein metabolism | 4-6 month pr patient

SECONDARY OUTCOMES:
Testosterone influence on Body composition by DEXA scan, Energy expenditure by indirect Calorimetry and VO2 max test | 4-6 month pr patient

CONTACTS AND LOCATIONS:
Overall Officials: Jens S Christensen, Professor, Principal Investigator — Medical Department M, Aarhus University Hospital, Denmark
Locations (1):
- Medical department M and Investigational Laboratories, Aarhus C, Jutland, Denmark

REFERENCES:
- [Background] Malkin CJ, Pugh PJ, Jones RD, Kapoor D, Channer KS, Jones TH. The effect of testosterone replacement on endogenous inflammatory cytokines and lipid profiles in hypogonadal men. J Clin Endocrinol Metab. 2004 Jul;89(7):3313-8. doi: 10.1210/jc.2003-031069. PMID 15240608
- [Derived] Host C, Gormsen LC, Christensen B, Jessen N, Hougaard DM, Christiansen JS, Pedersen SB, Jensen MD, Nielsen S, Gravholt CH. Independent effects of testosterone on lipid oxidation and VLDL-TG production: a randomized, double-blind, placebo-controlled, crossover study. Diabetes. 2013 May;62(5):1409-16. doi: 10.2337/db12-0440. Epub 2012 Nov 27. PMID 23193189